CLINICAL TRIAL: NCT00951483
Title: Cardiovascular Biomarkers During Quetiapine Treatment of Depression
Brief Title: Cardiovascular Biomarkers and Quetiapine in Depression and Anxiety Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Angelos Halaris, Professor, Loyola University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201880
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Depression; Anxiety
Keywords: Cardiovascular Biomarkers; Depression; Quetiapine
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Cohort (Experimental): Patients will undergo baseline psychological and laboratory tests then receive Quetiapine-XR(Seroquel-XR) with flexible dosing at the discretion of the treating physician based on clinical response and tolerability. The dose range will be from 50-300mg. The total duration of the treatment will be 12 weeks.
  Interventions: Drug: Quetiapine-XR
- Healthy Control (No Intervention): Participants without major depressive disorder or anxiety are enrolled as a comparison group without intervention.

INTERVENTIONS:
Drug: Quetiapine-XR — Quetiapine-XR (Seroquel-XR) 50-300mg daily for 12 weeks.
  Other Names: Seroquel
  Arms: Intervention Cohort

SUMMARY:
No suitable treatment has been identified to reverse and ideally prevent, the cardiovascular disease risk associated with depression and anxiety. The purpose of this study is to determine if quetiapine treatment of depression can reverse the signs of arterial stiffening that often occurs in depression and anxiety, and which are believed to be risk factors for future heart disease.

DETAILED DESCRIPTION:
The evidence that depressive and anxiety disorders confer a high relative risk (RR) for cardiovascular disease (CVD) development is clear and compelling. A cadre of inflammation, platelet activation and other biomarkers of endothelial dysfunction strongly suggest multiple and possibly interrelated mechanisms underlying this co-morbidity. Early detection of the vulnerability to develop CVD has become an urgent health issue. However, detection alone of vulnerability without proper therapeutic intervention aimed at reversing it, is merely of scientific interest. The evidence to date that antidepressant drugs, while highly efficacious in restoring euthymia, may not normalize the biomarkers of CVD vulnerability. Hence, there is a need to identify other pharmacologic interventions for depression. Quetiapine, due to its unique molecular structure and unique pharmacological profile, belongs to none of the known classes of antidepressants. However, quetiapine clearly has antidepressant and anti-anxiety efficacies. Now, we propose to explore whether quetiapine can reverse those pathophysiological changes occurring in mixed depression/anxiety that have been linked causally to the development of CVD. Accordingly, the primary purpose of this study is to compare C-Reactive Protein between the treatment and healthy control groups at 12 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Major Depressive Disorder (MDD), first episode or recurrent, by Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) requiring treatment. The index episode must be at least 14 days of persistent symptoms. If first episode, patients must not have been previously treated. If recurrent, must not be receiving treatment for the recurrence.
* Females and males 20-65 years of age
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at time of enrolment
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Females who are pregnant, lactating, breast feeding or on oral contraceptives
* Any DSM-IV Axis I disorder not defined in the inclusion criteria except MDD co-morbid with generalized anxiety disorder (GAD)
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine (Seroquel) as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Concomitant use of any other antidepressant, anxiolytic, or antipsychotic agent
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before the study begins
* Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* History of heavy smoking within the preceding 6 months
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
* Restrictions prior to blood drawings: Aspirin (previous 240 hours), antihistamines (previous 72 hours), Tylenol (previous 72 hours), Vitamin C or E (previous 72 hours), sleeping pills (previous 72 hours), caffeinated beverages (8 hours), physical exertion (8 hours) and tobacco products (2 hours).
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrolment in the present study.
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%.
  * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
  * Not under physician care for DM
  * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
  * Physician responsible for patient's DM care has not approved patient's participation in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelos Halaris, MD, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Health System, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-one individuals were consented and 47 participants received study drug while 44 participants enrolled as healthy control participants between July 2009 and October 2011. Participants were recruited using physician solicitation and advertisements.
Groups:
- Healthy Control: Participants without major depressive disorder or anxiety are enrolled as a comparison group without intervention. They will undergo baseline psychological and laboratory tests and will be followed for 12 weeks.
Period: Overall Study
Arm/Group | Intervention Cohort | Healthy Control
Started | 47 | 44
Completed | 28 | 44
Not Completed | 19 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 15 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis were conducted on all individuals who signed an informed consent document (N = 91)
Groups:
- Experimental Cohort: Patients will undergo baseline psychological and laboratory tests then receive Quetiapine-XR(Seroquel-XR) with flexible dosing at the discretion of the treating physician based on clinical response and tolerability. The dose range will be from 50-300mg. The total duration of the treatment will be 12 weeks.
  Quetiapine-XR: Quetiapine-XR (Seroquel-XR) 50-300mg daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental Cohort | Healthy Control | Total
Number analyzed (Participants) | 47 | 44 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.1) | 39.5 (13.8) | 41.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 21 | 15 | 36
Race/Ethnicity, Customized [Number; unit: Participants]
  Non-Hispanic White | 22 | 30 | 52
  African American | 13 | 8 | 21
  Asian | 1 | 3 | 4
  Hispanic White | 11 | 3 | 14
Tobacco Use [Number; unit: Participants]
  Non-Smoker | 22 | 40 | 62
  Smoker | 0 | 3 | 3
  Unknown | 25 | 1 | 26
Height [Mean (Standard Deviation); unit: Meters] — Height was measured in meters
  Meters | 1.66 (0.19) | 1.68 (0.10) | 1.67 (0.15)
Weight [Mean (Standard Deviation); unit: kilograms] — Weight was measured in kilograms
  kilograms | 88.50 (23.8) | 74.59 (15.45) | 81.86 (21.31)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.98 (6.76) | 26.51 (5.77) | 29.36 (6.84)
Menopausal Status [Number; unit: participants]
  Premenopausal | 23 | 19 | 42
  Postmenopausal | 3 | 10 | 13
  Not Applicable (Males) | 21 | 15 | 36
Family History of Depression [Number; unit: participants]
  No | 17 | 38 | 55
  Yes | 22 | 2 | 24
  Unknown | 8 | 4 | 12
Concomitant Psychiatric Medication [Number; unit: participants]
  Yes | 26 | 1 | 27
  No | 16 | 42 | 58
  Unknown | 5 | 1 | 6
Family History of Alzheimer's Disease [Number; unit: participants]
  No | 18 | 36 | 54
  Yes | 21 | 4 | 25
  Unknown | 8 | 4 | 12
Baseline Hamilton Rating Scale for Depression with Seven Items [Median (Inter-Quartile Range); unit: units on a scale] — The seven item Hamilton Rating Scale for Depression (HAMD-7) is an objective assessment of depression administered by a trained rater. This version allows scores to range from 0 to 22, where higher scores indicate worsening mood.
  units on a scale | 15 [13 to 19] | 0 [0 to 1] | 8 [0 to 15]
Baseline Hamilton Rating Scale for Depression with 17 Items [Median (Inter-Quartile Range); unit: units on a scale] — The 17-item Hamilton Rating Scale for Depression (HAMD-17) is an objective assessment of depression administered by a trained rater. This version allows scores to range from 0 to 52, where higher scores indicate worsening mood.
  units on a scale | 25 [20 to 29] | 0 [0 to 2] | 17 [0 to 25]
Baseline Hamilton Rating Scale for Depression with 21 Items [Median (Inter-Quartile Range); unit: units on a scale] — The 21-item Hamilton Rating Scale for Depression (HAMD-21) is an objective assessment of depression administered by a trained rater. This version allows scores to range from 0 to 63, where higher scores indicate worsening mood.
  units on a scale | 27 [23 to 32] | 0 [0 to 2] | 18 [0 to 27]
Baseline Hamilton Rating Scale for Anxiety [Median (Inter-Quartile Range); unit: units on a scale] — The 14-item Hamilton Rating Scale for Anxiety (HAM-A) is an objective assessment of anxiety administered by a trained rater. This version allows scores to range from 0 to 56, where higher scores indicate worsening anxiety.
  units on a scale | 22 [15 to 28] | 0 [0 to 1] | 10 [0 to 22]
Baseline Beck Depression Inventory [Median (Inter-Quartile Range); unit: units on a scale] — The 21-item Beck Depression Inventory (BDI) is a subjective self-report assessment of depression. This version allows scores to range from 0 to 63, where higher scores indicate worsening mood.
  units on a scale | 25.50 [17.75 to 33.50] | 0 [0 to 1.25] | 16.50 [1.00 to 28.75]
Perceived Stress Scale with 14 Items [Median (Inter-Quartile Range); unit: units on a scale] — The 14-item Perceived Stress Scale (PSS-14) is a subjective self-report assessment of stress. Each item is rated on a five point frequency scale ranging from 0 = never experiencing the stress symptom to 4 = Very often experiencing the stress symptom. Scores range from 0 to 56, where higher scores indicate higher stress.
  units on a scale | 49.50 [44.25 to 54.00] | 27.00 [24.00 to 32.00] | 43.50 [30.50 to 52.00]

OUTCOME MEASURES:

1. Primary Outcome: C-Reactive Protein at 12 Weeks
Description: To compare C-Reactive Protein between the treatment and healthy control groups at 12 weeks post treatment.
Time Frame: 12 weeks
Population: Due to the cost for the C-reactive protein assay, only 20 individuals from each cohort are analyzed (N = 40).
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Experimental Cohort | Healthy Control
Number analyzed (Participants) | 20 | 20
mg/L | 3.31 [1.06 to 8.21] | 0.50 [0.30 to 2.4]
Statistical Analysis 1: Comparison: Experimental Cohort vs Healthy Control; The null hypothesis is that C-reactive protein (CRP) is no different between the experimental and healthy control cohorts at 12 weeks; Test type: Superiority or Other; p = .001, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -2.65

2. Secondary Outcome: Change in Hamilton Rating Scale for Depression With Seven Items (HAM-D-7)
Description: The seven item Hamilton Rating Scale for Depression (HAMD-7) is an objective assessment of depression administered by a trained rater. This version allows scores to range from 0 to 22, where higher scores indicate worsening mood.
Time Frame: Baseline and 12 weeks
Population: This analysis is restricted to the twenty-eight individuals from the intervention cohort who had valid HAM-D-7 responses at baseline and 12 weeks; the healthy control arm is not included here, because their HAM-D-7 scores were recorded at baseline only (see baseline characteristics).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Intervention Cohort Baseline; Intervention Cohort End of Treatment: Patients will undergo baseline psychological and laboratory tests then receive Quetiapine-XR(Seroquel-XR) with flexible dosing at the discretion of the treating physician based on clinical response and tolerability. The dose range will be from 50-300mg. The total duration of the treatment will be 12 weeks.
  Quetiapine-XR: Quetiapine-XR (Seroquel-XR) 50-300mg daily for 12 weeks.
Arm/Group | Intervention Cohort Baseline | Intervention Cohort End of Treatment
Number analyzed (Participants) | 28 | 28
units on a scale | 15.00 [12.25 to 19.75] | 3.00 [0.00 to 10.75]
Statistical Analysis 1: Comparison: Intervention Cohort Baseline vs Intervention Cohort End of Treatment; The null hypothesis is that there is no difference between the intervention cohort's baseline HAM-D-7 score and end of treatment (i.e., 12 week) HAM-D-7 score; Test type: Superiority or Other; p < .001, Wilcoxon signed rank test; z-score = -4.544

3. Secondary Outcome: Change in Hamilton Rating Scale for Depression With 17 Items (HAM-D-17)
Description: The 17-item Hamilton Rating Scale for Depression (HAMD-17) is an objective assessment of depression administered by a trained rater. This version allows scores to range from 0 to 52, where higher scores indicate worsening mood.
Time Frame: Baseline and 12 weeks
Population: This analysis is restricted to the twenty-eight individuals from the intervention cohort who had valid HAM-D-17 responses at baseline and 12 weeks; the healthy control arm is not included, because their HAM-D-17 scores were recorded at baseline only (see baseline characteristics).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Cohort Baseline | Intervention Cohort End of Treatment
Number analyzed (Participants) | 28 | 28
units on a scale | 24.00 [20.00 to 28.75] | 5.50 [1.00 to 14.75]
Statistical Analysis 1: Comparison: Intervention Cohort Baseline vs Intervention Cohort End of Treatment; The null hypothesis is that there is no difference between the intervention cohort's baseline HAMD-17 score and end of treatment (i.e., 12 week) HAMD-17 score; Test type: Superiority or Other; p < .001, Wilcoxon signed rank test; z-score = -4.627

4. Secondary Outcome: Change in Hamilton Rating Scale for Depression With 21 Items (HAMD-21)
Description: The 21-item Hamilton Rating Scale for Depression (HAMD-21) is an objective assessment of depression administered by a trained rater. This version allows scores to range from 0 to 52, where higher scores indicate worsening mood.
Time Frame: Baseline and 12 weeks
Population: This analysis is restricted to the twenty-eight individuals from the intervention cohort had valid HAM-D-21 responses at baseline and 12 weeks; the healthy control arm is not included, because their HAM-D-21 scores were recorded at baseline only (see baseline characteristics).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Cohort Baseline | Intervention Cohort End of Treatment
Number analyzed (Participants) | 28 | 28
units on a scale | 26.50 [22.50 to 32.00] | 6.50 [1.25 to 16.75]
Statistical Analysis 1: Comparison: Intervention Cohort Baseline vs Intervention Cohort End of Treatment; The null hypothesis is that there is no difference between the intervention cohort's baseline HAMD-21 score and end of treatment (i.e., 12 week) HAMD-21 score; Test type: Superiority or Other; p < .001, Wilcoxon signed rank test; z-score = -4.624

5. Secondary Outcome: Change in Hamilton Rating Scale for Anxiety (HAM-A)
Description: The 14-item Hamilton Rating Scale for Anxiety (HAM-A) is an objective assessment of anxiety administered by a trained rater. This version allows scores to range from 0 to 56, where higher scores indicate worsening anxiety.
Time Frame: Baseline and 12 weeks
Population: This analysis is restricted to the twenty-eight individuals from the intervention cohort had valid HAM-A responses at baseline and 12 weeks; the healthy control arm is not included, because their HAM-A scores were recorded at baseline only (see baseline characteristics).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Cohort Baseline | Intervention Cohort End of Treatment
Number analyzed (Participants) | 28 | 28
units on a scale | 22.00 [15.25 to 28.00] | 6.00 [1.25 to 10.00]
Statistical Analysis 1: Comparison: Intervention Cohort Baseline vs Intervention Cohort End of Treatment; The null hypothesis is that there is no difference between the intervention cohort's baseline HAM-A score and end of treatment (i.e., 12 week) HAM-A score; Test type: Superiority or Other; p < .001, Wilcoxon signed rank test; z-score = -4.510

6. Secondary Outcome: Change in Beck Depression Inventory (BDI)
Description: The 21-item Beck Depression Inventory (BDI) is a subjective self-report assessment of depression. This version allows scores to range from 0 to 63, where higher scores indicate worsening mood.
Time Frame: Baseline and 12 weeks
Population: This analysis is restricted to the twenty-seven individuals from the intervention cohort had valid BDI responses at baseline and 12 weeks; the healthy control arm is not included, because their BDI scores were recorded at baseline only (see baseline characteristics).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Cohort Baseline | Intervention Cohort End of Treatment
Number analyzed (Participants) | 27 | 27
units on a scale | 25.00 [17.00 to 33.00] | 6.00 [1.00 to 18.00]
Statistical Analysis 1: Comparison: Intervention Cohort Baseline vs Intervention Cohort End of Treatment; The null hypothesis is that there is no difference between the intervention cohort's baseline BDI score and end of treatment (i.e., 12 week) BDI score; Test type: Superiority or Other; p < .001, Wilcoxon signed rank test; z-score = -4.435

7. Secondary Outcome: Change in 14-item Perceived Stress Scale (PSS-14)
Description: The 14-item Perceived Stress Scale (PSS-14) is a subjective self-report assessment of stress. Each item is rated on a five point frequency scale ranging from 0 = never experiencing the stress symptom to 4 = Very often experiencing the stress symptom. Scores range from 0 to 56, where higher scores indicate higher stress.
Time Frame: Baseline and 12 weeks
Population: This analysis is restricted to the twenty-three individuals from the intervention cohort had valid PSS-14 responses at baseline and 12 weeks; the healthy control arm is not included, because their PSS-14 scores were recorded at baseline only (see baseline characteristics).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Cohort Baseline | Intervention Cohort End of Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | 50.00 [43.00 to 54.00] | 35.00 [26.00 to 44.00]
Statistical Analysis 1: Comparison: Intervention Cohort Baseline vs Intervention Cohort End of Treatment; The null hypothesis is that there is no difference between the intervention cohort's baseline PSS-14 score and end of treatment (i.e., 12 week) PSS-14 score; Test type: Superiority or Other; p < .001, Wilcoxon signed rank test; z-score = -3.911

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 12 Week trial.
Arm/Group | Experimental Cohort | Healthy Control
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/44
Other Adverse Events (participants affected / at risk) | 39/47 | 0/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Cohort (N=47) | Healthy Control (N=44)
Weight gain (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 6 (6) | 0 (0)
Insomnia (General disorders) | 3 (3) | 0 (0)
Drowsiness (General disorders) | 10 (10) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 13 (13) | 0 (0)
Increased appetite (General disorders) | 5 (5) | 0 (0)
Increased irritability (General disorders) | 5 (5) | 0 (0)
Increased anxiety (Psychiatric disorders) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No